CLINICAL TRIAL: NCT00226317
Title: Phase 4 Study: An Open Prospective Study of the Safety and Effectiveness of Aripiprazole in the Treatment of Bipolar Depression
Brief Title: Aripiprazole in the Treatment of Bipolar Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cambridge Health Alliance (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHA-IRB-0030/01/04
Record Dates: First submitted 2005-09-12; First posted 2005-09-27 (Estimated); Last update posted 2017-04-18 (Actual); Status verified 2017-04

CONDITIONS: Bipolar Disorder
MeSH Terms: conditions — Bipolar Disorder | interventions — Aripiprazole

STUDY DESIGN:
Oversight: FDA-regulated Device: No

ARMS (1):
- Aripiprazole in depression treatment (Experimental)
  Interventions: Drug: Aripiprazole

INTERVENTIONS:
Drug: Aripiprazole

SUMMARY:
A systematic open-label prospective pilot study to assess aripirazole for acute bipolar depression, with a secondary assessment of longer-term mood stabilization.

DETAILED DESCRIPTION:
Study is 6 weeks long with 7 clinical visits.

ELIGIBILITY:
Inclusion Criteria:

* DSM-IV diagnosis of bipolar disorder, any subtype; MADRS >16; MRS < 10; not currently taking other mood stabilizers; women of reproductive potential must use an acceptable method of birth control

Exclusion Criteria:

* Current substance abuse within past month; serious unstable medical condition; active suicidal ideation; pregnant, trying to become pregnant, or nursing; intent to continue or initiate herbal preparations

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2004-04; Primary Completion 2007-12 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
Depression state | 6 week study

CONTACTS AND LOCATIONS:
Overall Officials: Robert T Dunn, MD, PhD, Principal Investigator — Cambridge Health Alliance
Locations (1):
- Cambridge Health Alliance, Cambridge, Massachusetts, United States